CLINICAL TRIAL: NCT00863603
Title: Artery Wall Hypoxia and Intimal Hyperplasia
Brief Title: The Effect of Oxygen on Healing an Artery From the "Injury" of Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical changes: graft to fistula first; enrollment of 46/132 planned. NIH approved animal model: supplemental oxygen/AV fistula.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0010M69621; R01HL076316 (NIH)
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: End Stage Renal Disease
Keywords: Supplemental oxygen; Intimal hyperplasia; Graft patency
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): No exposure to supplemental oxygen
- Oxygen, treatment, supplement (Other): 6 weeks of supplemental oxygen delivered by nasal cannula post hemodialysis graft placement
  Interventions: Other: oxygen

INTERVENTIONS:
Other: oxygen — 5 Liter/minute by nasal cannula for 6 wks
  Arms: Oxygen, treatment, supplement

SUMMARY:
Many grafts placed for dialysis access fail which causes patients to undergo additional operations, decreases their quality of life, and increases health care costs. The purpose of this study is to see if dialysis access grafts will function longer for patients who receive additional oxygen by means of a nasal cannula for 42 days after placement of their graft.

Patients will have periodic blood tests to measure oxygen levels in their blood. A series of ultrasound examinations of patient's dialysis grafts will be taken to ensure the graft is open and to measure the cellular proliferation (intimal hyperplasia) for comparison in those receiving extra oxygen and those with no oxygen.

DETAILED DESCRIPTION:
Vascular bypass grafting is a commonly performed procedure in vascular and cardiovascular surgery and the preferred bypass grafts are autogenous vein. Creation of a vascular anastomosis (AVA) is required at 2 sites (proximal and distal anastomoses) for every synthetic bypass graft. It is estimated that 50% of vascular bypass failures are due to anastomotic intimal hyperplasia (AIH). Intimal thickening of the artery wall is a normal response to healing at an anastomosis. Progression of intimal thickening leads to a pathological, hyperplastic, occlusive lesion - AIH, which in turn results in myocardial infarction, stroke, limb loss, death, graft failure, repeat operative procedures, and increased medical costs.

Our laboratory demonstrated in a rabbit model of AIH that: 1) there is a significant decrease in the delivery of oxygen to the peri-anastomotic artery wall following creation of a prosthetic vascular graft to artery anastomosis, 2) the oxygen gradient across the artery wall in the area of a prosthetic vascular graft anastomosis normalizes over a period of 6 weeks as healing occurs, 3) the gradient can be normalized immediately following an anastomosis by the administration of supplemental oxygen, and 4) the amount of AIH and smooth muscle cell proliferation can be reduced by immediately administering supplemental oxygen following creation of the anastomosis.

The long-range goal of our program is to understand the role of oxygen in blood vessel wall pathology. The specific objective of this project, which is the next step in the pursuit of our long-range program goal, is to determine if supplemental oxygen can inhibit AIH in a human graft model.

METHODS: Following review of inclusion and exclusion criteria suitable patients undergo surgical placement of a graft for hemodialysis. Following surgery, patients randomized to oxygen will breathe 5L supplemental oxygen during waking hours for 42 days. Periodic ultrasounds will be taken to assess graft function and patency and to measure intimal thickness. Patients will be followed for two years or until their graft fails.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80+/- referred and considered a candidate for a synthetic hemodialysis access graft.
2. Baseline room air arterial blood concentration >70 and arterial carbon dioxide concentration 45 mmHg. Pulmonary function tests > 75% predicted values
3. Currently undergoing dialysis
4. No previous synthetic hemodialysis grafts placed in the same arm (fistula in ipsilateral arm permitted)
5. Ability to use 5L/minute supplemental oxygen by nasal cannula
6. Nonsmoker, able to avoid other situations which would constitute a risk for use of oxygen
7. Medical condition with > 1 year life expectancy
8. Currently on no medications which would interfere with wound healing (i.e. steroids, chemotherapeutic agents)
9. Not pregnant nor planning to become pregnant during study period

Exclusion Criteria:

1. Failure to meet inclusion criteria
2. Failure to comply with study protocol for 3 consecutive days during the 6 wk oxygen/non-oxygen supplement period immediately following graft placement
3. Medical condition developing during study period causing a significantly worsening pulmonary function requiring supplemental oxygen for > 3 days
4. Need to take medication during study period which would interfere with wound healing any time during the 6 week period immediately following graft placement or need to take chronic medications (> 6 weeks) during the remainder of the study period.
5. Patient desire to withdraw
6. Failure of evidence of adequate increase in arterial blood oxygen concentration (pa02 > 115 for oxygen supplemented and pa02 > 55 mmHg for control obtained from arterial access port during dialysis run
7. Failure to use supplemental oxygen (if in supplemental oxygen group) at least 18 hours per day (as recorded in journal) -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The effect of supplemental oxygen on intimal thickness at the site of a hemodialysis access graft | Assessing intimal thickness in the first 2 yrs after graft placement

SECONDARY OUTCOMES:
Compare graft patency in oxygen supplemented vs. non oxygen supplemented group | Assessing graft patency in the first two years after graft placement

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Santilli, MD, PhD, MBA, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Veterans Affairs Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Division of Vascular Surgery, Minneapolis, Minnesota

REFERENCES:
- [Background] Tretinyak AS, Lee ES, Uema KM, d'Audiffret AC, Caldwell MP, Santilli SM. Supplemental oxygen reduces intimal hyperplasia after intraarterial stenting in the rabbit. J Vasc Surg. 2002 May;35(5):982-7. doi: 10.1067/mva.2002.123090. PMID 12021715
- [Background] Santilli SM, Wernsing SE, Lee ES. The effect of supplemental oxygen on the transarterial wall oxygen gradients at a prosthetic vascular graft to artery anastomosis in the rabbit. Ann Vasc Surg. 2001 Jul;15(4):435-42. doi: 10.1007/s100160010119. PMID 11525533
- [Background] Lee ES, Caldwell MP, Tretinyak AS, Santilli SM. Supplemental oxygen controls cellular proliferation and anastomotic intimal hyperplasia at a vascular graft-to-artery anastomosis in the rabbit. J Vasc Surg. 2001 Mar;33(3):608-13. doi: 10.1067/mva.2001.113495. PMID 11241134
- [Background] Santilli SM, Tretinyak AS, Lee ES. Transarterial wall oxygen gradients at the deployment site of an intra-arterial stent in the rabbit. Am J Physiol Heart Circ Physiol. 2000 Oct;279(4):H1518-25. doi: 10.1152/ajpheart.2000.279.4.H1518. PMID 11009436
- [Background] Santilli SM, Wernsing SE, Lee ES. Transarterial wall oxygen gradients at a prosthetic vascular graft to artery anastomosis in the rabbit. J Vasc Surg. 2000 Jun;31(6):1229-39. doi: 10.1067/mva.2000.104590. PMID 10842160
- [Background] Lee ES, Bauer GE, Caldwell MP, Santilli SM. Association of artery wall hypoxia and cellular proliferation at a vascular anastomosis. J Surg Res. 2000 Jun 1;91(1):32-7. doi: 10.1006/jsre.2000.5891. PMID 10816346
- [Background] Santilli SM, Kronson J, Payne WD. The effect of hypercholesterolemia on the rabbit transarterial wall oxygen gradient. Ann Vasc Surg. 1998 Sep;12(5):418-23. doi: 10.1007/s100169900178. PMID 9732418
- [Background] Santilli SM, Kronson JW, Payne WD. Cigarette smoking alters the rabbit transarterial wall oxygen gradient. Ann Vasc Surg. 1998 Mar;12(2):174-81. doi: 10.1007/s100169900137. PMID 9514238
- [Background] Santilli SM, Stevens RB, Anderson JG, Caldwell MD. The effect of aging on the transarterial wall oxygen gradient. Ann Vasc Surg. 1995 Mar;9(2):146-51. doi: 10.1007/BF02139656. PMID 7786699
- [Background] Santilli SM, Stevens RB, Anderson JG, Payne WD, Caldwell MD. Transarterial wall oxygen gradients at the dog carotid bifurcation. Am J Physiol. 1995 Jan;268(1 Pt 2):H155-61. doi: 10.1152/ajpheart.1995.268.1.H155. PMID 7840259
- [Background] Santilli SM, Fiegel VD, Knighton DR. Alloxan diabetes alters the rabbit transarterial wall oxygen gradient. J Vasc Surg. 1993 Aug;18(2):227-33. PMID 8350431
- [Background] Santilli SM, Fiegel VD, Knighton DR. Changes in the aortic wall oxygen tensions of hypertensive rabbits. Hypertension and aortic wall oxygen. Hypertension. 1992 Jan;19(1):33-9. doi: 10.1161/01.hyp.19.1.33. PMID 1730436
- [Background] Santilli SM, Fiegel VD, Aldridge DE, Knighton DR. Rabbit aortic endothelial cell hypoxia induces secretion of transforming growth factor beta and augments macrophage adhesion in vitro. Ann Vasc Surg. 1991 Sep;5(5):429-38. doi: 10.1007/BF02133047. PMID 1958457